CLINICAL TRIAL: NCT03734549
Title: Predicting Procedural and Long-term Outcomes of Endovascular Revascularization for Lower Extremity Peripheral Artery Chronic Total Occlusions With Computed Tomographic Angiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTUAF2017LSK-137
Record Dates: First submitted 2018-06-26; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-06

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- technical success group: Technical success was defined as crossing the CTO and placement of a guidewire in the distal true lumen confirmed by angiography.
- technical failure group: Technical failure was defined that guidewire could not crossing through the CTO nor reture to the true lumen by angiography.
- had adverse events group: Patients had one of the adverse events such as all-cause death, nonfatal myocardial infarction, repeat revascularization or amputation.at 12 months after procedures.
- had no adverse events group: Patients had none adverse events such as all-cause death, nonfatal myocardial infarction, repeat revascularization and amputation at 12 months after procedures

SUMMARY:
Nearly one-half of all lower extremity percutaneous interventions performed in patients with symptomatic peripheral artery disease (PAD) involve chronic total occlusions (CTOs) which are technically more challenging and are associated with more periprocedural complications and lower rates of procedural success comparing with non CTOs. Despite innovate dedicated CTO devices developed and provides higher technical success, a wire-catheter approach to cross peripheral artery CTO is most often the first choice of operators as its lower cost advantage.Subhash Banerjee MD reported of all 1,362 CTOs, wire-catheter approaches were used in 82% and the technical success rate was 65%. If the operators chose wire-catheter as primary crossing device at the beginning of the procedure, but the technically failed with the provisional use of re-entry or crossing devices to try to procedural success. Such procedures add incrementally to procedure duration and cost and the revascularization and amputation rate at 12 month were highly increased comparing with using dedicated CTO devices initially. So it is very important to predict the outcome of guidewire crossing through CTOs to direct the choice of crossing strategy.

Current data suggested that computed tomography angiography (CTA) imaging of PAD and a detailed comprehensive assessment for CTO arteries before endovascular therapy can assist preprocedural planning to maximize procedural success. Previous studies about coronary CTOs prediction scores as the KCCT score and CT-based CT-RECTOR provide the factors including occlusion length, the shape of proximal entry site, severe calcification, and etc. characters base on CTA correlating with the outcome of cross. As the same physiopathologic mechanism, we hypothesized that the radiographic characteristics are connected with outcomes of guidewire crossing occlusions. To our knowledge, few studies focused on how to predict the successful GC through peripheral artery CTO, therefore, the purpose of this study was to establish a simple and clinically applicable prediction model based on CTA characters within the occlusive lesions and clinical parameters to predict the GC outcomes of patients with lower extremity CTO.

In addition, the long-term effect of endovascular revascularization are very important. An analysis concluded that limb adverse event (repeat revascularization rate 17.2%, amputation rates 8.5%) at 12-month in the CTOs with direct wire-catheter crossing strategy. Base on the proven influence factors (the lesion length, small diameter of the vessel and severe calcification, mechanical exposure, etc.)of adverse event at after endovascular revascularization ,we also can establish model with preoperative computer tomography angiography that provided the lesion detail characteristic combing the patients' biochemical and clinical feature to predict the adverse event rate at 12-month after endovascular revascularization.

DETAILED DESCRIPTION:
Patients Patients with peripheral artery disease met the inclusion criteria if they were PAD patients, had performed preprocedural CTA and PTA. The hospital's database was used to identify the patients met inclusion criteria. The medical records and radiologic information system database were reviewed to retrieve clinical information including background diseases and radiographic findings.

Computed Tomography Angiography Protocol A 128-section multidetector CT (Philips brillianceiCT was used for scanning with the following scanning parameters，tube voltage was 120 kVp, tube current 40-440mA, and 0.625-mm slice thicknesses. The protocols required patients to lie supine with legs extended, A fixed bolus of contrast medium with total volume of 90 ml (370 mg iodine per milliliter) was injected into antecubital vein at a rate of 4 mL/sec, followed by a 30 mL saline flush, by using a dual-barrel power injector. CT scanning was performed with the coverage from the common iliac artery bifurcation to the tiptoe. Scanning began 12 seconds after an attenuation threshold of 150 HU was reached.

CTA Data Analysis CTA data were transferred to an offline workstation for further analysis. Axial images, cross-sectional views, curved planar reformations (CPR), and multiplanar reformations (MPR), as well as three-dimensional maximum intensity projection images were available for evaluation. We measure the degree of transluminal calcification, CT attenuation value of the proximal occlusion ,anatomic distribution of the leision,and length of occlusion,and the degree of stenosis CTO Crossing Strategy CTO crossing strategy was wire-catheter. Technical success was defined as crossing the CTO and placement of a guidewire in the distal true lumen confirmed by angiography.Outcomes include binary variables of lesion crossing described as technical success or failure.

Follow-up We also examined patient adverse events after procedures at 12 months: all-cause death,nonfatal myocardial infarction,revascularization and amputation.

Built prediction model we can establish model with preoperative computer tomography angiography that provided the lesion detail characteristic combing the patients' biochemical and clinical feature to predict the procedural and long-term outcomes of endovascular revascularization for Lower extremity peripheral artery chronic total occlusions.

ELIGIBILITY:
Inclusion Criteria:

* PAD patients with CTOs confirmed by angiograpy underwent pre-procedue CTA and endovascular revascularization

Exclusion Criteria:

* Patients' clinical date were incomplete; The interval between preprocedural CTA and PTA. was more than one month The CTA images could not be evaluated because of motion and metal artifact Loss to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAD patients with CTOs confirmed by angiograpy underwent pre-procedue CTA and endovascular revascularization
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
technical success | At time of procedure (day 0)
  Successful crossing the CTO and placement of a guidewire in the distal true lumen confirmed by angiography

SECONDARY OUTCOMES:
Composite of Major Adverse Events | 12 months
  the incidence of major adverse events (composite of all-cause death, nonfatal myocardial infarction, repeat revascularization or amputation) during the 12-month study period

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, archiater, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China